CLINICAL TRIAL: NCT06108479
Title: A Phase I/Ib, First-In-Human, Multi-Part, Open-Label Study to Investigate the Safety, Tolerability, Pharmacokinetics, Biological and Clinical Activity of DF6215 Monotherapy and in Combination Therapy in Patients with Advanced (Unresectable, Recurrent, or Metastatic) Solid Tumors
Brief Title: Study of DF6215 in Patients with Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dragonfly Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DF6215-001; KEYNOTE-G13 (Other: Merck); MK-3475-G13 (Other: Merck)
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor, Adult; Solid Tumor Cancer
Keywords: DF6215-001; DF6215; Melanoma; HPV-Positive Advanced Malignancies; Ovarian Cancer; Head and Neck Cancer; Non-Small Cell Lung Cancer; Renal Cell Carcinoma; Advanced or Metastatic Solid Tumors; Antineoplastic Agents; Antineoplastic Agents, Immunological; Molecular Mechanisms of Pharmacological Action; Neoplasms; Solid Tumor; Dose Escalation; oncology; pembrolizumab; KEYTRUDA®
MeSH Terms: conditions — Melanoma; Ovarian Neoplasms; Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Monotherapy Dose Escalation (Experimental): Patients will receive DF6215 monotherapy, with dose levels escalated to determine the MTD of DF6215 monotherapy.
  Interventions: Drug: DF6215
- Combination Therapy Dose Escalation (Experimental): Patients will receive DF6215 in combination with pembrolizumab to determine the MTD of DF6215 in combination with pembrolizumab.
  Interventions: Drug: DF6215; Drug: pembrolizumab; Drug: KEYTRUDA®
- Monotherapy Dose Enrichment (Experimental): Patients with advanced melanoma after prior anti-PD-1 treatment will receive DF6215 monotherapy at two different dose levels to further characterize the doses selected during the Dose Escalation (monotherapy) part.
  Interventions: Drug: DF6215
- Monotherapy Expansion of DF6215 in Advanced Melanoma (Experimental): Patients with advanced melanoma after prior anti-PD-1 will receive DF6215 monotherapy at the recommended efficacy expansion dose to evaluate the clinical activity of DF6215 in monotherapy.
  Interventions: Drug: DF6215
- Combination Expansion of DF6215 and pembrolizumab in PROC (Experimental): Patients with platinum-resistant ovarian cancer (PROC) will receive DF6215 in combination with pembrolizumab at the recommended efficacy expansion dose to evaluate the clinical activity of DF6215 in combination with pembrolizumab.
  Interventions: Drug: DF6215; Drug: pembrolizumab; Drug: KEYTRUDA®
- Combination Expansion of DF6215 and pembrolizumab in Advanced Melanoma (Experimental): Patients with advanced melanoma after prior anti-PD-1 therapy will receive DF6215 in combination with pembrolizumab at the recommended combination efficacy expansion dose to evaluate the clinical activity of DF6215 in combination with pembrolizumab.
  Interventions: Drug: DF6215; Drug: pembrolizumab; Drug: KEYTRUDA®
- Monotherapy Expansion of DF6215 in Multiple Tumor Types (Basket) (Experimental): Patients with multiple tumor types will receive DF6215 monotherapy at the recommended efficacy expansion dose to evaluate the clinical activity of DF6215 in monotherapy.
  Interventions: Drug: DF6215
- Combination Expansion of DF6215 and pembrolizumab in Multiple Tumor Types (Experimental): Patients with multiple tumor types will receive DF6215 in combination with pembrolizumab at the recommended combination efficacy expansion dose to evaluate the clinical activity of DF6215 in combination with pembrolizumab.
  Interventions: Drug: DF6215; Drug: pembrolizumab; Drug: KEYTRUDA®
- DF6215 Monotherapy Safety/PK/PD (Experimental): Expansion cohorts of DF6215 in multiple dose levels after evaluation for safety in the DF6215 Dose Escalation arm. Additional Pharmacokinetic (PK) and Pharmacodynamic (PD) samples included in this arm.
  Interventions: Drug: DF6215

INTERVENTIONS:
Drug: DF6215 — Immunotherapy (cytokine) targeting effector cells.
Drug: pembrolizumab — Anti-PD-1 immunotherapy agent
  Arms: Combination Expansion of DF6215 and pembrolizumab in Advanced Melanoma; Combination Expansion of DF6215 and pembrolizumab in Multiple Tumor Types; Combination Expansion of DF6215 and pembrolizumab in PROC; Combination Therapy Dose Escalation
Drug: KEYTRUDA® — Anti-PD-1 immunotherapy agent
  Arms: Combination Expansion of DF6215 and pembrolizumab in Advanced Melanoma; Combination Expansion of DF6215 and pembrolizumab in Multiple Tumor Types; Combination Expansion of DF6215 and pembrolizumab in PROC; Combination Therapy Dose Escalation

SUMMARY:
A Phase I/Ib, First-In-Human, Multi-Part, Open-Label Study to Investigate the Safety, Tolerability, Pharmacokinetics, Biological and Clinical Activity of DF6215 Monotherapy and in Combination Therapy in Patients with Advanced (Unresectable, Recurrent, or Metastatic) Solid Tumors; is designed to assess the safety, tolerability, and preliminary efficacy of DF6215 alone or in combination with pembrolizumab in patients with advanced solid tumors. The study is open-label, meaning both participants and investigators are aware of the treatment being administered.

DETAILED DESCRIPTION:
This Phase I/Ib trial involves multiple parts and includes both dose-escalation and dose-expansion phases. The primary objectives are to evaluate the safety and tolerability of DF6215, an investigational biologic agent, when administered either as a monotherapy or in combination with pembrolizumab, a known immunotherapy drug, and evaluate the clinical activity of DF6215 monotherapy and in combination with pembrolizumab. Secondary objectives include assessing pharmacokinetics, pharmacodynamics, and preliminary efficacy based on tumor response using RECIST 1.1 criteria. The trial will enroll adult patients with advanced (unresectable, recurrent, or metastatic) solid tumors, and the study design allows for dose modifications based on safety monitoring and the occurrence of dose-limiting toxicities (DLTs). The trial will also incorporate a safety monitoring committee to review data at regular intervals to ensure patient safety .

ELIGIBILITY:
Key Inclusion Criteria

* Male or female patients ≥ 18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* An estimated life expectancy of ≥ 3 months.
* Adequate hematological function.
* Normal pulmonary function.
* Adequate hepatic function.
* Adequate renal function.
* Effective Contraception.
* Additional Inclusion Criteria apply to each cohort.

Key Exclusion Criteria

* Patients receiving chemotherapy, radiotherapy (other than palliative bone-directed radiotherapy), major surgery, or receiving another systemic anticancer therapeutic agent within 28 days before the start of study drug(s) or within 5 half-lives of the previous therapeutic agent (if known), whichever is shorter.
* Patients receiving any of the following concurrent anticancer treatments or investigational drugs within 28 days before the start of the study drug(s), or within 5 half-lives of the previous therapeutic agent (if known), whichever is shorter:

  * Cytoreductive therapy
  * Radiotherapy (except for palliative bone-directed radiotherapy)
  * Note: ≤ 2 weeks of palliative radiotherapy for non-CNS disease is permitted. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study drug.
  * Immune therapy
  * Cytokine therapy (except for erythropoietin)
  * Major surgery (excluding prior diagnostic biopsy)
  * Concurrent systemic therapy with steroids or other immunosuppressive agents.
  * Note that short-term administration of systemic steroids (eg, for allergic reactions or the management of irAEs) and physiologic dose steroids (≤ 10 mg prednisone, or equivalent) for those with treated brain metastases are allowed. Patients receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug(s) will be excluded.
  * Bisphosphonate or denosumab initiated within 14 days of the first dose of study drug(s)
* Previous malignant disease, other than the target malignancies to be investigated in this study, within the last 3 years. Exceptions (eg, basal or squamous cell carcinoma of the skin, low grade prostate cancer [Gleason score ≤ 6 and must be Stage I or II], or cervical carcinoma in situ) may be considered on a case-by-case basis, in consultation with the Medical Monitor.
* Any of the following cardiac abnormalities:

  * A clinically relevant abnormality on the electrocardiogram (ECG)
  * Clinically relevant coronary artery disease (CAD) or uncontrolled congestive heart failure
  * Medically uncontrolled angina pectoris
  * An implantable pacemaker or automatic implantable cardioverter-defibrillator
  * A history of risk factors for ventricular tachycardia, torsades de pointes, fainting, unexplained loss of consciousness, or convulsions
  * A history of heart failure, congestive heart failure, cardiomyopathy, uncontrolled hypokalemia, hypomagnesemia, or hypoglycemia; any evidence of conduction abnormality (eg, increased QRS complex)
  * Congenital long QT syndrome or a prolonged QTc mean on screening ECG
  * QTc > 470 msec for women and > 450 msec for men
  * History of myocardial infarction within 6 months before the first dose of study drug(s)
  * Received sotalol within 10 days of the first dose of study drug(s), or received a medication known to prolong the ECG QT interval within 14 days of the first dose of study drug(s)
  * A heart rate of < 50 or > 100 bpm at rest on screening ECG
* Patients aged more than 50 years must have a normal cardiac stress test.
* Patients with history of CAD must have a normal stress test (eg, thallium or technetium-99m sestamibi) and be cleared to participate in the study.
* History of ocular/uveal melanoma or mucosal melanoma.
* Primary tumor site of nasopharynx (any histology).
* Patients with brain metastases are excluded, unless all of the following criteria are met:

  * CNS lesions are asymptomatic and previously treated
  * Patient does not require ongoing daily steroid treatment for replacement for adrenal insufficiency (except ≤ 10 mg prednisone [or equivalent]) for at least 14 days before the first dose of study drug
  * Imaging demonstrates stable disease 28 days after last treatment
* Receipt of any organ transplant, including autologous or allogeneic stem-cell transplantation.
* Patients must not have received aldesleukin or any other experimental IL-2 based drug, including intralesional administration.
* Significant acute or chronic hepatitis B virus (HBV), hepatitis C virus (HCV) infection during the screening window, as well as historic positive for human immunodeficiency virus (HIV) or clinically significant active infections that render the patient ineligible for study treatment as determined by the treating investigator.

  * Patients with known HIV infection are excluded unless they meet the following criteria:
  * Must have CD4+ T-cell (CD4+) counts ≥ 350 cells/μL at the time of screening, and
  * Must have no history of AIDS-related opportunistic infections of HIV-associated conditions such as Kaposi sarcoma or multicentric Castleman's disease, and
  * Patients on antiretroviral therapy (ART) must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 or the LLOQ (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks before screening and agree to continue ART throughout the study
* Preexisting autoimmune disease (except vitiligo) needing treatment with systemic immunosuppressive agents for more than 28 days within the last 3 years, or clinically relevant immunodeficiencies (eg, dysgammaglobulinemia or congenital immunodeficiencies). Patients with a history of immune related endocrinopathies (eg, hypothyroidism, hyperthyroidism, and type 1 diabetes mellitus) that are stable on hormone replacement therapy are eligible for this study.
* Patients with a known medical history of keratitis, ulcerative keratitis, or corneal perforation.
* Patients with known history of neurologic conditions, cerebrovascular accident, or seizures.
* Known severe hypersensitivity reactions to mAbs (≥ Grade 3 as defined by NCI-CTCAE v5.0), any history of anaphylaxis, or uncontrolled asthma (ie, 3 or more features of partly controlled asthma).
* Persisting toxicity related to a prior therapeutic agent > Grade 1 as defined by NCI CTCAE v5.0 (however, ≤ Grade 2 alopecia, ≤ Grade 2 endocrinopathies, and ≤ Grade 2 sensory neuropathy are acceptable).
* Patients in certain cohorts with prior anti-PD-1 and anti-PD-L1 treatment are eligible for the study, unless they have experienced any of the following:

  * Grade 3 or 4 treatment-related toxicity during an anti-PD-1 or anti-PD-L1 treatment (excluding Grade 3 or 4 immune-related endocrinopathies adequately controlled with hormone replacement therapy).
  * Grade 2 treatment-related toxicity that impacted either the lungs, the nervous system, or the cardiac system, during an anti-PD-1 or anti-PD-L1 treatment (patients with a history of Grade 2 peripheral neuropathy, or paresthesia, not related to anti-PD-1 or anti-PD-L1 treatments are eligible).
  * For combination basket cohorts: received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
  * For combination basket cohorts: received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher irAE (except endocrine disorders that can be treated with replacement therapy) or was discontinued from that treatment due to Grade 2 myocarditis or recurrent Grade 2 pneumonitis.
* Known alcohol or drug abuse.
* Severe dyspnea at rest due to complications of advanced malignancy.
* Requiring supplementary oxygen therapy.
* All other significant diseases (eg, inflammatory bowel disease) which, in the opinion of the Investigator, might impair the patient's ability to participate.
* Legal incapacity or limited legal capacity.
* Unable to understand or give signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in the protocol. Examples include certain psychiatric conditions.
* Patients who have received a live or live-attenuated vaccine within 30 days before the first dose of study drug. Administration of killed vaccines is allowed.
* Pregnant or lactating.
* Severe hypersensitivity (≥ Grade 3) to study drugs and/or any of their excipients.
* Additional Exclusion Criteria apply to each cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of DF6215 Monotherapy and in Combination with Pembrolizumab | First 28 days for monotherapy; first 42 days for combination therapy.
  Determine the maximum tolerated dose of DF6215 both as monotherapy and when combined with pembrolizumab, by assessing the occurrence of dose-limiting toxicities.
Safety and Tolerability of DF6215 Monotherapy and in Combination with Pembrolizumab | Continuously throughout the study, up to 2 years.
  Evaluate the safety and tolerability of DF6215 monotherapy and in combination with pembrolizumab at various dose levels by monitoring the incidence, severity, and causality of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs), and TEAEs leading to discontinuation, per Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Efficacy Expansion: Clinical Activity of DF6215 monotherapy and in combination of Pembrolizumab | Assessed from the start of treatment until disease progression or study end, up to 2 years.
  To evaluate the clinical activity of DF6215 monotherapy and in combination with pembrolizumab, measured by ORR per investigator assessment as defined by RECIST 1.1 in the efficacy expansion part.

SECONDARY OUTCOMES:
Clinical Activity: Objective Response Rate (ORR), Disease Control Rate (DCR), and Clinical Benefit Rate (CBR) | Assessed every 8 weeks until disease progression or study termination, up to 2 years.
  Evaluate the clinical activity of DF6215 monotherapy and in combination with pembrolizumab, measured by ORR, DCR, and CBR as per RECIST 1.1.
Pharmacokinetics (PK) Parameters | Samples collected at predetermined time points across the first and second cycles and periodically thereafter.
  Assess the PK of DF6215 monotherapy and in combination with pembrolizumab at multiple dose levels, measured by PK parameters such as area under the concentration-time curve (AUC0-t), maximum concentration (Cmax), minimum concentration (Cmin), time to reach maximum concentration (tmax), and half-life (t½).
Immunogenicity: Incidence of Anti-Drug Antibodies (ADAs) | Samples collected at predetermined time points across the first and second cycles and periodically thereafter.
  To assess the immunogenicity of DF6215 monotherapy and in combination with pembrolizumab, measured by incidence of patients with anti-drug antibodies against DF6215.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (9):
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - University of California San Diego Moores Cancer Center, San Diego, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Tampa General Hospital, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - NYU Langone Health, New York, New York
  - Lifespan - Rhode Island Hospital, Providence, Rhode Island
  - SCRI Oncology Partners, Nashville, Tennessee
- Australia (2):
  - Cancer Research SA (CRSA), Adelaide, South Australia
  - Peninsula and South East Oncology Medical (PASO), Frankston, Victoria
- France (10):
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - CHU de Marseille - Hôpital de la Timone, Marseille
  - Institut Paoli-Calmettes, Marseille
  - Institut Curie, Paris
  - Hôpital Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Institut de Cancérologie de l'Ouest - Saint-Herblain - Site René Gauducheau, Saint-Herblain
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse

IPD SHARING:
Plan to Share IPD: No